CLINICAL TRIAL: NCT06738238
Title: To Compare Effects of Eldova Technique and Corrective Exercises in Upper Cross Syndrome
Brief Title: Comparative Effects of Eldova Technique and Corrective Exercises in Upper Cross Syndrome
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Riphah/RCRAHS/REC/MS-PT/09136
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Upper Cross Syndrome
Keywords: Upper cross syndrome; ELDOA; Corrective exercises
MeSH Terms: conditions — Oculocerebral hypopigmentation syndrome type Preus

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eldova (Experimental): Elongation Longitudinaux Avec Decoaption Osteo Articulaire
  Interventions: Other: ELDOA
- Corrective exercises (Experimental): corrective exercises
  Interventions: Other: ELDOA; Other: CORRECTIVE EXERCISES

INTERVENTIONS:
Other: ELDOA — In this, each position will be maintained for 1 minute Level: C0/C1/C2 The patient is side lying with bottom arm folded under the head and maintain the neck in a horizontal position with the spine. the bottom leg is bent to stabilize the torso in a vertical position.
  Level: C4/C5 Patient lying in supine position and raise both hand arm towards the roof of the room with extended wrist. Bilateral knee to chest with planter flexion at ankle joint.
  Level: C5/C6 Same position as for c4/c5 with the arms will be elevated 120 degree Level C6/C7 Supine position with one arm abducted 90 degree and wrist joint at extension and the other hand abducted 30degrees with wrist joint at extension and one leg knee to chest and one leg raise with knee extension and planter flexion at ankle joint.
  Level: T4/T5 Quadruped position with one arm abducted 90degrees with wrist at extension Level: T6/T7. Conventional TX is Hot Pack, Tens for 10min. Patient is assessed through baseline, week 1, week 2 and week 4.
Other: CORRECTIVE EXERCISES — All position will be held for 10 seconds. Initial phase Duration of this phase is 2 weeks. Exercise 1: lying supine on a foam roll with different abduction angles Exercise 2: side lying with external rotation Exercise 3: side lying with forward flexion Exercise 4: standing diagonal flexion Exercise 5: military press Improvement phase. Duration of this phase is 1 week we only add thera- band and dumbbells to the previously mentioned exercises Exercise 1: side lying external rotation with dumbbell Exercise 2: side lying forward flexion with dumbbell Exercise 3: standing diagonal flexion with thera-band Exercise 4: standing external rotation with thera band. Exercise 5: abduction in sitting on training ball. Exercise 6: lying prone on foam ball with different abduction angles Maintenance phase. Duration of this phase is 1 week. Conventional treatment Hot Pack, Tens for 10 minutes Patient is assessed through baseline, week 1, week 2 and week 4.
  Arms: Corrective exercises

SUMMARY:
The objective of the study is to compare the effects of ELDOA technique and corrective exercises in Upper cross syndrome. The study will be randomized control trial including two experimental groups having 42 participants in each group.

DETAILED DESCRIPTION:
Musculoskeletal disorders are most common among people aged between 20 to 50 years with primary complaint of headache and neck pain due to their abnormal posture for prolong time. Upper cross syndrome refers to a specific muscles imbalance in upper quadrant of the body. Which brings postural deviation and may affects cervicothoracic and glenohumeral joints movements.Upper cross syndrome alters muscle activation pattern in the neck, trunk and scapula muscles and affect movement pattern of scapula along with postural deviation. These abnormalities lead to various musculoskeletal symptoms in the upper body.Upper cross syndrome is also referred as cervical cross syndrome is described as predictive pattern of alternative tightness and weakness of upper traps, pectoralis muscles, leavator scapulae, rhomboid, and serratus anterior and deep flexors of the neck. These muscles changes also alter the stability of glenohumeral joint stability which end up in more abduction due to the tightness of levator scapulae muscle.Due to the weakness of serratus anterior muscle, which affect the stability of scapula and alter the movement pattern of the scapula than lead to scapular dyskinesia.Scapular dyskinesia is a term that refers to, the alteration in the function and position of scapula. Scapular dyskinesis is further divided in two separates groups, static scapular positional(the asymmetry in the scapular resting position which can be observed by looking to the scapula in which inferior border is prominent and dynamic scapular stability (the alteration in the scapular motion with arm alleviation due alteration in scapular stabilizer muscles). The clinical assessment of scapula have three methods (A) direct observation (Lateral scapular slide test,(B) manually assisted movements(scapular assistance test),(C) assessment of surrounding structures. Scapula dyskinesia can be treated by stretching of the tight muscles and strengthening of the weak muscles. As mention earlier weakness of lower trap, med trap, serratus anterior and tightness of upper trap, pects muscles and levator scapulae occur with upper cross syndrome which can lead to scapula alteration, rounded shoulder and forward head posture. Due to abnormal posture of cervical in upper cross syndrome can cause forward head syndrome . Hyperextension of upper cervical(C1/C2) and hyper flexion of lower cervical (C3-C7) is referred to Forward head posture. Many studies have been conducted regarding treatment of upper cross syndrome through stretching and strengthening but the gap in previous literature is that there is no study designed yet to evaluate and compare both eldova technique and corrective exercises. Current study had addressed the comparison of eldova technique and corrective exercises in upper cross syndrome with the aim of evaluating and identifying the most effective intervention for managing this specific condition, the integration of Eldova techniques and corrective exercises in Upper cross syndrome management offers a holistic approach that addresses both structural and functional aspects, aiming for optimal outcomes in pain relief, postural correction, and functional restoration.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female subjects
* Age between 15 to 35 years
* Subjects with scapular dyskinesia
* Subject with rounded shoulders

Exclusion Criteria:

* Subjects with cervical discogenic pain
* Subjects with spinal stenosis
* Cervical spine surgery

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-12-13 (Estimated); Study Completion 2024-12-13 (Estimated)

PRIMARY OUTCOMES:
Lateral scapular slide test. | 4 weeks
  The scapular position is measured by taking the side to side differences between both sides in all 3 test positions. The measurements are taken from the inferior angle of the scapulae to the spinous process of the thoracic vertebrae on horizontal plane. The test is done in 3 positions, with the arm abducted to 0, 45 and 90 degrees in the coronal plane.
  Position 1 involves placing the shoulder in neutral position, with the arms relaxed at the sides, Position 2 the humerus is placed in medial rotation and 45degree abduction, by positioning patients hands around the waist, Position 3 the humerus is placed in maximal rotation and 90degree abduction.
  The Test is positive when there is a difference of 1.5 cm when measurements are compared bilaterally.
Forward head posture (tragus to wall) | 4 weeks
  Horizontal distance between tragus of the ear and wall, standing with heels and buttocks against the wall (to prevent pivoting), knees extended and chin. Nine and half centimeter is normal anything greater than this value indicate FHP.
Neck pain | 4 weeks
  is strongly associated with upper body dysfunction and can affect daily lives activities. To measure neck pain before and after treatment neck disability index questionnaire will be filled from participant's neck disability index questionnaire with score of more than 20%.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Mudassir Shah, MS-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Madina colony, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Treatment of Upper Crossed Syndrome: A Narrative Systematic Review — https://pubmed.ncbi.nlm.nih.gov/37628525/